CLINICAL TRIAL: NCT04244318
Title: Randomized Clinical Trial to Evaluate the Results of the ODISEA-T Model, in a Sample of Fathers, Mothers and/or Caregivers and Children and Adolescents Belonging to AFT Programs of La Protectora de la Infancia, Chile.
Brief Title: ODISEA Trauma: Parental Therapy Dispositive + Videofeedback 3.0
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esteban Gómez Muzzio (Other)
Responsible Party: Sponsor-Investigator, Esteban Gómez Muzzio, Phd, Executive Director, Fundacion America por la Infancia
Organization: Fundacion America por la Infancia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCT:ODISEA-T
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Parent-Child Relations; Parenting; Parent-child Problem
Keywords: video feedback intervention; randomized controlled trial; parenting skills; ODISEA; video-feedback; parental therapy; parental trauma; complex trauma
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Masking Description: Due to the characteristics of the intervention and the allocation, neither caregivers nor the professionals will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- G1: DTP + Videofeedback 3.0 (Experimental): Once a week, it will be offered a 5-session intervention of parental therapy (DTP). After that, a 5-session intervention of videofeedback.
  Parental Therapy. S1: the therapist will talk with caregiver about her childhood and attachment figures. S2: family mandates and how they have influenced his life. S3: integration of painful memories and the "inner child". S4: focus on the present time, and rearing. S5: exploring expectations and stimulating a commimment to positive parenting.
  Videofeedback. S1: a play interaction between the child and the caregiver will be recorded for 10 minutes. S2: will be done between the therapist and caregivers, where they will watch different selected parts of the video and will provide feedback through a mentalization constructed framework. S3: another play interaction video will be recorded, that will be discussed on the S4 with the caregiver. S5: a final interaction video will be recorded.
  Interventions: Behavioral: Video-feedback ODISEA 3.0; Behavioral: ODISEA-DTP: parental therapy
- G2: Videofeedback 3.0 + DTP (Experimental): Once a week, it will be offered a 5-session intervention of videofeedback. After that, a 5-session intervention of parental therapy (DTP).
  Videofeedback. S1: a play interaction between the child and the caregiver will be recorded for 10 minutes. S2: will be done between the therapist and caregivers, where they will watch different selected parts of the video and will provide feedback through a mentalization constructed framework. S3: another play interaction video will be recorded, that will be discussed on the S4 with the caregiver. S5: a final interaction video will be recorded.
  Parental Therapy. S1: the therapist will talk with caregiver about her childhood and attachment figures. S2: family mandates and how they have influenced his life. S3: integration of painful memories and the "inner child". S4: focus on the present time, and rearing. S5: exploring expectations and stimulating a commimment to positive parenting.
  Interventions: Behavioral: Video-feedback ODISEA 3.0; Behavioral: ODISEA-DTP: parental therapy
- Control Group (Active Comparator): Patients in control group will be placed as an active comparator group, as "treatment as usual" due to the nature of the psychosocial program from wich the cases were selected. After collecting the post-test data, they will be offered the same intervention than the experimental group.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Video-feedback ODISEA 3.0 — Video-feedback intervention ODISEA 3.0 (Gómez & Maureira, 2022), which incorporates an attachment theory framework. This intervention was constructed within the ODISEA's comprehensive and formative model of parenthood which was developed in Chile by Dr. Esteban Gómez Muzzio (Gómez, 2022).
  Other Names: videofeedback
  Arms: G1: DTP + Videofeedback 3.0; G2: Videofeedback 3.0 + DTP
Behavioral: ODISEA-DTP: parental therapy — Parental Therapy (ODISEA-DTP, Gómez & Maureira, 2022): is a parental therapy strategy that works over 5 sessions with the history of caregivers in a systematic way, allowing to explore their past, present and expected future concerning parenting, child rearing, attachment and child abuse, between other issues. The DTP is a protocolized model of parental therapy, each session is carefully designed to elicit memories, emotions and to stimulate reflective function (about the past and their own childhood) and parental reflective function (about the present with the child).
  Other Names: Parental Therapy
  Arms: G1: DTP + Videofeedback 3.0; G2: Videofeedback 3.0 + DTP
Behavioral: Treatment as usual — Psychosocial intervention (parental education, family counseling, home visits and school and Court coordination) for child abuse and neglect, implemented by six Family Therapeutic Programs (AFT) of the NGO "Protectora de la Infancia"
  Arms: Control Group

SUMMARY:
This is a study protocol of a randomized controlled trial, which aims to validate the effectiveness of the ODISEA Trauma intervention (parental thearpy + videofeedback) compared to a control group. The data collection will be through a three point evaluation (pre, medium and post intervention) using the parenting skills questionnaire (E2P short form), parental stress index - short form (PSI-SF), the adult emotional regulation questionnaire (ERQ), an adult reflective function questionnaire, the parental reflective function questionnaire (PRFQ), the child abuse potential inventory (CAPI), and the socioemotional competence scale for children (ECOS). Additionally, caregivers will be screened for ACES and with a sociodemographic characterization questionnaire. At the same time, profesionals will be assessing caregivers using an scale to measure complex trauma in adults (ECTA). The primary outcome aims to measure the effectiveness of the intervention within the parenting domain (positive parenting practices) and parental trauma (complex trauma, adult emotion regulation, reflective function and child abuse potential of the caregivers). The secondary outcomes will be to assess parenting stress, socioemotional competencies of children and implementation fidelity compared to accumulated risk.

DETAILED DESCRIPTION:
This research is designed as a randomized controlled trial, with 1:1 allocation ratio. The randomization will be performed through block randomization. The participating sites for this study will be 6 family therapeutic programas of ONG "Protectora de la Infancia" in Chile, where the trained professionals are currently working.

1. Specific objectives.

   The primary objective of this research is to determinate the effectiveness of the ODISEA Trauma Intervention (ODISEA-T) in improving parental resilience, strengthening parenting skills and reducing child abuse potential controlled by parental trauma, accumulated risk and parenting stress in caregivers of children aged 0 to 17 years of age, compared to the control group.

   Furthermore, the key secondary objectives are the following:
   1. To measure the effect of ODISEA-T on the pre-post evaluation of parental resilience through the symtoms scale of the adult complex trauma ECTA scale.
   2. To measure the effect of ODISEA-T on a pre-post evaluation of the positive parenting practices using the short form of the E2P scale.
   3. To measure the effect of ODISEA-T on a pre-post evaluation of child abuse potential using the CAPI.
   4. To measure the effect of ODISEA-T on a pre-post evaluation of adult emotion regulation using the ERQ.
   5. To measure the effect of ODISEA-T on a pre-post evaluation of reflective function of caregivers using the RFQ.
   6. To measure the effect of ODISEA-T on a pre-post evaluation of parental reflective function of caregivers using the PRFQ.
   7. To measure the effect of ODISEA-T on a pre-post evaluation of parenting stress levels through the PSI-SF parental stress index - short form.
   8. To measure the effect of ODISEA-T on a pre-post evaluation of children socioemotional competencies through the ECOS scale.
   9. And lastly, to explore the relationship between intervention fidelity and accumulated risk (ACES) and complex trauma (ECTA full scale).
2. Intervention.

Eligible caregivers will be randomized in equal ratio, between three posible conditions: (a) "treatment as usual" control group; (b) ODISEA-T intervention group 1; and (c) ODISEA-T intervention group 2.

The model ODISEA-T consist of a combined 5 sessions of Parental Therapy (ODISEA-DTP: parental therapeutic dispositive) and 5 sessions of Videofeedback (Videofeedback ODISEA 3.0).

* The ODISEA-T intervention group 1 will offer parental therapy followed by videofeedback.
* The ODISEA-T intervention group 2 will offer videofeedback followed by parental therapy.
* The control group, after five months "treatment as usual" intervention, will receive ODISEA-T either way as an ethical consideration.

The ODISEA-DTP: parental therapeutic dispositive (Gómez & Maureira, 2022) is a parental therapy strategy that works over 5 sessions with the history of caregivers in a systematic way, allowing to explore their past, present and expected future concerning parenting, child rearing, attachment and child abuse, between other issues. The DTP is a protocolized model of parental therapy, each session is carefully designed to elicit memories, emotions and to stimulate reflective function (about the past and their own childhood) and parental reflective function (about the present with the child).

The Video-feedback ODISEA 3.0 (Gómez & Maureira, 2022) strategy is sequenced in three moments, a) a video recording of the caregiver-child dyad interaction, b) the selection of specific 10-20 seconds interactions sequences which are later discussed by the professional in charge of the dyad, and c) a feedback and reflective process guided by the professional with the caregiver. In this research, the basic five-session Video-feedback ODISEA 3.0 model will be implemented, consisting of (1) a game session recorded on video between the caregiver and the child, (2) followed by a reflective session between the professional and the caregiver, which will be guided using different segments of the video, concentrating on the resources of the caregivers, (3) succeeded by the second recorded game session between the caregiver and the child, (4) continuing with a second reflective session between the caregiver and the professional, integrating more challenging aspects of the interaction, (5) concluding with the last recorded video session of the dyad.

All families assigned to the control group will receive the intervention five months after the pre-test as an ethical decision. Therefore, the comparator will be set as treatment as usual, because all families are participating of a social program focused on cases fo child maltreatment (and cannot be without any kind of intervention).

Considering the counterfactual deliberations from this methodology, for instance the differentiation between the specific's intervention -ODISEA-T- influence against common elements such as the professional's empathy, warmth, listening skills, among others, this elements will be embedded and assessed through a thoughtful fidelity criteria evaluation of the implementation process in order to differentiate the treatment's contributions.

For a given caregiver, the intervention may be needed to be discontinued by the researchers for reasons of withdrawal of the participant consent. Even though there are no risks associated to this intervention, in a rare case of withdrawal because of emotional damage, this will be considered as an adverse event and a protocol has been constructed for managing this situation.

For managing the co-intervention bias, every caregiver will be asked to complete different questions of other interventions that they be considered as concomitant care in addition to the parental therapy + video-feedback intervention that may impact on this trial, such as parenting schools, psychotherapy, among others.

After gathering the sample, an external professional from the NGO "Protectora de la Infancia" will send the folios (not the names) of the cases, and then a research professional through a random numerical assignment will generate a block randomization for the dyads. Once assigned to the control group or experimental group 1 or experimental group 2, the dyads will be given a document that will reinforce what is explained in the informed consent, in informing in which group they been placed, and acknowledging that both groups will have the same intervention.

Due to the characteristics of the intervention and the allocation, neither caregivers nor the professionals will be blinded.

Pre-randomization information will be recorded, regarding the interested caregivers that did not meet all the inclusion criteria, for example not giving their consent. Post-randomization losses will also be recorded.

By August 2024 it is expected a sample of 215 participating dyads from 6 different social programs of NGO "Protectora de la Infancia". Participants will be identified and contacted by the intervention professional, having no relationship with the principal investigator. Their participation is voluntary and has no economic cost to them.

The sample will be recruited through 6 social programs of NGO "Protectora de la Infancia". There will be a participation agreement signed by the directors of the NGO institution participating in this study.

An external professional will proceed to generate the blocked randomization, using a random number generator. When a caregivers agree to participate in the study, the coordinator will give the data to this researcher who till inform the intervention professional the corresponding allocation. All caregivers who gives consent for the study and fulfil the inclusion criteria will be randomized. After the enrollment of each professional, the data will be requested by the study coordinator, which will be assigned to the external researcher to proceed to the randomization.

DATA ANALYSIS

Eight evaluation instruments (ECTA, E2P, CAPI, ERQ, RFQ, PRFQ, PSI-SF, ECOS) will be used as dependent variables.

* ANCOVA will be used to measure the effect of the intervention for each of the different evaluation instruments.
* To explore the relationship between the number of adverse experiences experienced in childhood and the fidelity of the treatment, as well as between complex trauma of the caregivers and the fidelity of treatment, a linear relationship measure between the two variables (simple regression) will be evaluated.
* Measure post-hoc data if the intervention has different effects on each of the dimensions of each instrument (post-hoc ANCOVA).

After proceeding with the data analysis, an outcome research paper will be provided for the scientific community.

DATA MANAGEMENT.

The intervention professionals will provide the gathered data to the research coordinator through two platforms, both password protected: The first platform is https://academia.americaporlainfancia.com/, a website designed to be used as a virtual classroom for the students of America por la Infancia. Therefore, it will be implemented a special section for researches, in which all the intervention professionals will have a username and password to access. In this platform, the different professionals will access the banner associated with this research - which only they can access with their user and personal and non-transferable passwords -, where they will enter the evaluation documents and family data. Only the research coordinator will be able to view and download the documents, and after downloading them they will be stored on the external hard drive that will be stored in the dependencies of Fundación América por la Infancia, being later eliminated from the virtual platform. The hard drive will remain in Los Filósofos 5029, commune of Macul, Santiago, Chile. The second platform is https://wetransfer.com/, a website on which, through the foundation's account, the professionals will send the videos to the coordinator's e-mail, videos that will be sent using a password. This platform allows sending large documents to emails. As the data, the videos will be downloaded, eliminated from the webpage, and stored on the same hard drive mentioned above.

A data monitoring committee (DMC) will not be necessary for this trial, because of the short durations and known minimal risks. Likewise, no interim analyses are considered for this study. Also, as this study is a multicenter trial, auditing will be considered both as an overall process, and for each recruiting center and their professionals, with the objective to monitor consents, completeness, adherence to the protocol, among other relevant data.

No ancillary studies are considered in the implementation of the study. If any tieried consent are constructed for future research unrelated to the this study and for different purposes form the main trial should be sent to the ethics committee and implemented in a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: Caregivers (≥ 18 years), with children between 1 month and 17 years.
* Sexes eligible for study: both.
* Accepts healthy volunteers: yes.
* Inclusion criteria for the adult: adult caregiver (≥ 18 years), mother, father or other caregiver of children between 1 month and 17 years
* Inclusion criteria for the child: Age between 1 month and 17 years.

Exclusion Criteria:

* Exclusion criteria for the adult: Court order which denies the adult to be with the child.
* Exclusion criteria for the child: No exclusion criteria.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference of the parental resilience | 5 months.
  Parental resilience is defined as a reduction of symptoms associated with complex trauma in the caregivers, assesed using a complex trauma scale in adults (ECTA).
Difference of the positive parenting practices | 5 months
  The perception or self-assessment that the adult has regarding their own parenting skills, which will be measured through the E2P short form positive parenting scale (Gómez, Contreras & Pezora, 2022). E2P is a self-report questionnaire that can be completed by any adult who has a caregiver role of a child between 0 and 17 years old.
Difference of child abuse potential | 5 months
  Child abuse potential concerns with the risk factors measured by using the Child Abuse Potential Inventory (CAPI, Milner).

SECONDARY OUTCOMES:
Difference of the adult emotion regulation | 5 months.
  Adult emotion regulation will be measured using the Emotion Regulation Questionnaire (ERQ).
Difference of the reflective function of caregivers | 5 months.
  Reflective function of caregivers will be measured using the Reflective Function Questionnaire (RFQ, Fonagy et al)
Difference of the parental reflective function of caregivers | 5 months.
  Parental Reflective Function of caregivers will be measured using the Parental Reflective Function Questionnaire (PRFQ, Fonagy et al)
Difference of parenting stress. | 5 months.
  Defined as a complex construct that combines characteristics of the caregivers, of the child and of the family, and how they interact to the person's evaluation of their role as caregiver (Abidin 1992, in Mc Kelvey et al 2008). Will be assessed through the PSI-SF.
Difference of children´s socioemotional competencies | 5 months.
  Socioemotional competencies of children (namely, socioemotional cognition, emotion regulation, and emotional communication, Gómez & Strasser, 2021) will be measured using the Socioemotional Competencies Scale (ECOS, Gómez & Strasser, 2023).
Difference of the fidelity of the intervention and its association with the accumulated risk of the caregivers. | 5 months.
  Accumulated risk was constructed incorporating the ACES (adverse childhood experiences) screening scale. By screening the adverse experiences that the caregiver had experienced in his or her childhood, it will be able to assign it in different complexity levels. According to the longitudinal study of adverse childhood experiences, 10 categories were defined that refer to high stress events that occur between 0 and 18 years of age (Felliti & Anda, 1998).
Difference of the fidelity of the intervention and its association with complex trauma of the caregivers. | 5 months
  Complex trauma of caregiver was constructed incorporating the ECTA scale. By evaluating the complex trauma indicators of caregivers, it will be able to assign it in different complexity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Gómez, Ph.D., Principal Investigator — Executive Director Fundación América por la Infancia
Locations (1):
- ONG Protectora de la Infancia, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bakermans-Kranenburg MJ, van IJzendoorn MH, Juffer F. Less is more: meta-analyses of sensitivity and attachment interventions in early childhood. Psychol Bull. 2003 Mar;129(2):195-215. doi: 10.1037/0033-2909.129.2.195. PMID 12696839
- [Background] Barone L, Barone V, Dellagiulia A, Lionetti F. Testing an Attachment-Based Parenting Intervention-VIPP-FC/A in Adoptive Families with Post-institutionalized Children: Do Maternal Sensitivity and Genetic Markers Count? Front Psychol. 2018 Feb 19;9:156. doi: 10.3389/fpsyg.2018.00156. eCollection 2018. PMID 29515483
- [Background] Cassidy J, Brett BE, Gross JT, Stern JA, Martin DR, Mohr JJ, Woodhouse SS. Circle of Security-Parenting: A randomized controlled trial in Head Start. Dev Psychopathol. 2017 May;29(2):651-673. doi: 10.1017/S0954579417000244. PMID 28401843
- [Background] Feder G, Ramsay J, Dunne D, Rose M, Arsene C, Norman R, Kuntze S, Spencer A, Bacchus L, Hague G, Warburton A, Taket A. How far does screening women for domestic (partner) violence in different health-care settings meet criteria for a screening programme? Systematic reviews of nine UK National Screening Committee criteria. Health Technol Assess. 2009 Mar;13(16):iii-iv, xi-xiii, 1-113, 137-347. doi: 10.3310/hta13160. PMID 19272272
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Finkelhor D. Screening for adverse childhood experiences (ACEs): Cautions and suggestions. Child Abuse Negl. 2018 Nov;85:174-179. doi: 10.1016/j.chiabu.2017.07.016. Epub 2017 Aug 4. PMID 28784309
- [Background] Fukkink RG. Video feedback in widescreen: a meta-analysis of family programs. Clin Psychol Rev. 2008 Jul;28(6):904-16. doi: 10.1016/j.cpr.2008.01.003. Epub 2008 Feb 5. PMID 18359136
- [Background] Juffer F, Struis E, Werner C, Bakermans-Kranenburg MJ. Effective preventive interventions to support parents of young children: Illustrations from the Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline (VIPP-SD). J Prev Interv Community. 2017 Jul-Sep;45(3):202-214. doi: 10.1080/10852352.2016.1198128. PMID 28641060
- [Background] Juffer F, Bakermans-Kranenburg MJ. Working with Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline (VIPP-SD): A case study. J Clin Psychol. 2018 Aug;74(8):1346-1357. doi: 10.1002/jclp.22645. Epub 2018 May 21. PMID 29781521
- [Background] Risholm Mothander P, Furmark C, Neander K. Adding "Circle of Security - Parenting" to treatment as usual in three Swedish infant mental health clinics. Effects on parents' internal representations and quality of parent-infant interaction. Scand J Psychol. 2018 Jun;59(3):262-272. doi: 10.1111/sjop.12419. Epub 2017 Dec 15. PMID 29244205
- [Background] Ramsauer B, Lotzin A, Muhlhan C, Romer G, Nolte T, Fonagy P, Powell B. A randomized controlled trial comparing Circle of Security Intervention and treatment as usual as interventions to increase attachment security in infants of mentally ill mothers: Study Protocol. BMC Psychiatry. 2014 Jan 30;14:24. doi: 10.1186/1471-244X-14-24. PMID 24476106
- [Background] Schoemaker NK, Jagersma G, Stoltenborgh M, Maras A, Vermeer HJ, Juffer F, Alink LRA. The effectiveness of Video-feedback Intervention to promote Positive Parenting for Foster Care (VIPP-FC): study protocol for a randomized controlled trial. BMC Psychol. 2018 Aug 3;6(1):38. doi: 10.1186/s40359-018-0246-z. PMID 30075813
- [Background] Suess GJ, Bohlen U, Carlson EA, Spangler G, Frumentia Maier M. Effectiveness of attachment based STEEP intervention in a German high-risk sample. Attach Hum Dev. 2016 Oct;18(5):443-60. doi: 10.1080/14616734.2016.1165265. Epub 2016 Apr 1. PMID 27035267
- [Background] Vilaseca R, Rivero M, Bersabe RM, Navarro-Pardo E, Cantero MJ, Ferrer F, Valls Vidal C, Innocenti MS, Roggman L. Spanish Validation of the PICCOLO (Parenting Interactions With Children: Checklist of Observations Linked to Outcomes). Front Psychol. 2019 Mar 27;10:680. doi: 10.3389/fpsyg.2019.00680. eCollection 2019. PMID 30971993
- [Background] West AL, Aparicio EM, Berlin LJ, Jones Harden B. IMPLEMENTING AN ATTACHMENT-BASED PARENTING INTERVENTION WITHIN HOME-BASED EARLY HEAD START: HOME-VISITORS' PERCEPTIONS AND EXPERIENCES. Infant Ment Health J. 2017 Jul;38(4):514-522. doi: 10.1002/imhj.21654. Epub 2017 Jun 30. PMID 28665540